CLINICAL TRIAL: NCT01848197
Title: An Open, Randomized, Parallel-group, Multicenter Clinical Study to Evaluate Efficacy and Safety of Paclitaxel Every 2 Weeks Compared Weekly in Adjuvant Treatment of Breast Cancer
Brief Title: Paclitaxol Every 2 Week Versus Paclitaxol Every 1 Week in the Adjuvant Treatment of Breast Cancer
Acronym: PATEN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taizhou Hospital (Other)
Responsible Party: Principal Investigator, Feilin Cao, MD, Taizhou Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZJTC0001
Record Dates: First submitted 2013-05-02; First posted 2013-05-07 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer; Paclitaxel; Epirubicin; Cyclophosphamide
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel

ARMS (2):
- EC-P2 (Experimental): all patients first received 4 cycles of intravenous epirubicin and cyclophosphamide at 3-week intervals and were then intravenous paclitaxel 2-week intervals for 4 cycles.
  Interventions: Drug: paclitaxel
- EC-P1 (Active Comparator): all patients first received 4 cycles of intravenous epirubicin and cyclophosphamide at 3-week intervals and were then intravenous paclitaxel 1-week intervals for 12 cycles.
  Interventions: Drug: paclitaxel

INTERVENTIONS:
Drug: paclitaxel

SUMMARY:
RATIONALE: Adjuvant chemotherapy has been proven to reduce significantly the risk for relapse and death in women with operable breast cancer.In the North American Inter-Group factorial trial design (CALGB 9741) the concept of dosedense adjuvant chemotherapy was further tested in patients with node-positive breast cancer.Weekly paclitaxel after standard adjuvant chemotherapy with epirubicin and cyclophosphamide improves disease-free and overall survival in women with breast cancer.Investigators asked if dose-dense 2-week intertreatment intervals (supported by the use of granulocyte-colony stimulating factor) were better than the conventional inconvenient weekly intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-70 years female operable breast cancer patients
2. Patients were required to register within 60 days from the final surgical procedure required to adequately treat the invasive primary tumor.
3. women who had operable,histologically confirmed adenocarcinoma of the breast with a. histologically involved positive lymph nodes b. or histologic diagnosis for three negative patients; c. or lymph node negative, HER2 positive(if HER2 + +, FISH (fluorescence in situ hybridization method)/CISH tests confirmed HER2 amplification is positive),but unable or intolerant to herceptin combined chemotherapy.
4. Karnofsky points greater than or equal to 70.
5. Postmenopausal women or HCG test results were negative, Women of child-bearing potential willing to use effective contraception during the study.
6. PATIENT CHARACTERISTICS:

Hematopoietic:

* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal
* TBIL no greater than 1.5 times upper limit of normal
* AKP no greater than 2.5 times upper limit of normal
* AST no greater than 2.5 times upper limit of normal
* ALT no greater than 2.5 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 times upper limit of normal

Cardiovascular:

* No history of myocardial infarction
* No congestive heart failure
* No significant ischemic or valvular heart disease

Other:

* No other prior invasive malignancies within the past 5 years except curatively treated basal or squamous cell skin cancer or carcinoma in situ of the cervix
* No hypersensitivity to paclitaxel or docetaxel or other similarly formulated drugs (with Cremophor or polysorbate)

Other protocol-defined inclusion/exclusion criteria may apply.

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2013-05; Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 3 years
  time from randomization to disease recurrence (including death from recurrence if it was the first manifestation of recurrence), death without recurrence, or contralateral breast cancer.

SECONDARY OUTCOMES:
disease-free survival | 5 years
  time from randomization to disease recurrence (including death from recurrence if it was the first manifestation of recurrence), death without recurrence, or contralateral breast cancer.
overall survival | 5 years
  time from randomization to disease death with/without recurrence breast cancer.

OTHER OUTCOMES:
Explore the relationship between neuropathy and DFS and the related predictive biomarkers (RWDD3 and TECTA gene SNP etc) | 3 years
Explore predictive biomarker of neutropenia; | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Feilin Cao, MD, Principal Investigator — Zhejiang Taizhou hospital